CLINICAL TRIAL: NCT04506502
Title: Functional Changes With Magnetic Muscle Stimulation of Abdominal Muscle
Brief Title: Functional Change With MMS
Acronym: FMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA19-003
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Results first posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Muscle Weakness
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Muscle Toning (Experimental): The treatments are designed to evaluate muscle toning, firming and strengthening in the abdomen.
  Interventions: Device: The ZELTIQ System

INTERVENTIONS:
Device: The ZELTIQ System — The MMS device will be used to perform the treatments.

SUMMARY:
Evaluate the safety and efficacy of magnetic muscle stimulation (MMS) of abdominal muscle.

ELIGIBILITY:
Inclusion Criteria

* Subject (healthy volunteer) has read and signed the study written informed consent form.
* Male or female ≥ 22 years and ≤65 years of age.
* Subject has not had weight change exceeding 5% of body weight in the preceding month.
* Subject agrees to maintain body weight within 5% during the study by not making any changes in diet or exercise routine during the course of the study.
* Subject has a BMI ≤ 30 as determined at screening.
* Subject agrees to have photographs taken of the treatment area(s) during the scheduled time periods.
* Subject agrees to refrain from any new abdominal muscle training exercises of the treatment area during the course of the study.

Exclusion Criteria

* Subject has had a recent surgical procedure(s) in the area of intended treatment and muscle contractions may disrupt the healing process.
* Subject needs to administer or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
* Subject has had an intrauterine contraceptive device inserted or removed within the past month.
* Subject has a bleeding disorder or hemorrhagic condition
* Subject is taking or has taken diet pills or supplements within the past month.
* Subject has an active implanted electrical device such as a cardiac pacemaker, cochlear implant, intrathecal pump, hearing aids, defibrillator, or drug delivery system.
* Subject has metal or electronic implants in or adjacent to the treatment area
* Subject has an abdominal hernia.
* Subject has pulmonary insufficiency.
* Subject has a cardiac disorder.
* Subject has a malignant tumor.
* Subject has been diagnosed with a seizure disorder such as epilepsy.
* Subject currently has a fever.
* Subject is diagnosed with Grave's disease.
* Subject has a growth plate in the treatment area
* Subject is pregnant or intending to become pregnant during the study period (in the next 9 months).
* Subject is lactating or has been lactating in the past 6 months.
* Subject is unable or unwilling to comply with the study requirements.
* Subject is currently enrolled in a clinical study of any unapproved investigational device, investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Any other condition or laboratory value that would, in the professional opinion of the Investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-07-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Innovation Research Center, Pleasanton, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per protocol, subjects received magnetic muscle stimulation (MMS) treatments in the abdominal area in 8 sessions over a 1-month period. Office follow-up visits were required at 4 days, 1 month, 2 months and 3 months after the final treatment. During all visits, subjects were assessed for pain and adverse events and required study activities were performed per protocol.
Groups:
- Magnetic Muscle Stimulation (MMS) Treatment Group: Each subject received two MMS treatment sessions, at least two days apart, per week for a four-week period. Treatment was performed on the abdominal region.
  The treatments are designed to evaluate muscle toning, firming and strengthening in the abdomen.
  The ZELTIQ System: The MMS device was used to perform the treatments.
Period: Overall Study
Arm/Group | Magnetic Muscle Stimulation (MMS) Treatment Group
Started | 16
Completed | 14
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Illness and subsequent quarantine requirements related to SARS-CoV-2 local guidelines | 1

BASELINE CHARACTERISTICS:
Population: Data presented here as planned and collected (all enrolled).
Arm/Group | Magnetic Muscle Stimulation (MMS) Treatment Group
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Satisfaction Questionnaire From Baseline to 1-month Post-Treatment Follow-up Visit
Description: Measurement of participant's perception about body shape, assessed using the Body Satisfaction Questionnaire (BSQ) at the 1-month post-treatment follow-up visit. The scale measures body image using a set of dichotomous items used to describe aspects of shape and appearance. The questionnaire has total score range from 10 to 50. An increase in score (when compared to baseline) reflects the participant's perceived improvement in appearance in the treated region (abdomen). Questionnaire results were tabulated as the numerical change between mean baseline scores and scores recorded at the 1-month post-treatment follow-up visit. A positive change reflects an increase in the body satisfaction questionnaire total score.
Time Frame: Baseline, 1-month post-treatment follow-up visit
Population: Two subjects were excluded from per protocol population due to incomplete treatments and withdrawal of consent. The Per Protocol population consisted of all treated subjects that received 8 MMS treatments and with a weight change of no more than 5% of total body weight at the time the 1-month assessments were performed compared to the weight obtained at the first treatment visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Magnetic Muscle Stimulation (MMS) Treatment Group
Number analyzed (Participants) | 14
units on a scale | 8.6 (5.4)

2. Primary Outcome: Number of Incidents of Device-Related Adverse Events
Description: The incidence of device-related adverse events (AE) including device-related serious AEs will be tabulated.
Time Frame: AE information will be collected from the time of enrollment to the final follow-up visit at 3-months following the final treatment (approximately 4 months).
Population: All participants enrolled in the study and treated with the EMS device were evaluated for adverse events throughout the study. Investigators determined if an AE was not related, possibly related, probably related or definitely related to the study device. Data is presented here as planned and collected per protocol by the total As-Treated Population (defined as all treated participants regardless of weight change).
Measure: Number; unit: Device-Related Adverse Events
Arm/Group | Magnetic Muscle Stimulation (MMS) Treatment Group
Number analyzed (Participants) | 16
Device-Related Adverse Events | 1

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of enrollment through the 4-week post final treatment follow-up visit, approximately 4 months.
Description: Safety data is presented here as planned and collected per protocol, by the total As-Treated Population (defined as all treated participants regardless of weight change).
Arm/Group | Magnetic Muscle Stimulation (MMS) Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 6/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magnetic Muscle Stimulation (MMS) Treatment Group (N=16)
Menstrual Cycle Irregularity (Reproductive system and breast disorders) | 1 (1)
Back Alignment Flare-up (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal Discomfort (Right Side) (General disorders) | 1 (1)
Upper Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cold (Virus) (General disorders) | 1 (1)
Tingling Sensation in Lower Leg (Right) (Nervous system disorders) | 1 (1)
Rash on Wrist (Right) (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/02/NCT04506502/Prot_SAP_001.pdf